CLINICAL TRIAL: NCT02869672
Title: Safety and Immunogenicity Study of ACYW135 Meningococcal Polysaccharide Vaccine Aged 2-50 Years Old
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Beijing Chaoyang District Centre for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: cycdc2016-5
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: ACYW135 Meningococcal Polysaccharide Vaccine
Keywords: safety; immunogenicity; vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- age of 18-50 years old, experimental (Experimental): 0.5 ml of Tiantan Biology ACYW135 meningococcal polysaccharide vaccine will be given.
  Interventions: Biological: Tiantan Biology ACYW135 meningococcal polysaccharide vaccine
- age of 18-50 years old, control (Active Comparator): 0.5 ml of Hualan Biology ACYW135 meningococcal polysaccharide vaccine will be given.
  Interventions: Biological: Hualan Biology ACYW135 meningococcal polysaccharide vaccine
- age of 7-17 years old,experimental (Experimental): 0.5 ml of Tiantan Biology ACYW135 meningococcal polysaccharide vaccine will be given.
  Interventions: Biological: Tiantan Biology ACYW135 meningococcal polysaccharide vaccine
- age of 7-17 years old, control (Active Comparator): 0.5 ml of Hualan Biology ACYW135 meningococcal polysaccharide vaccine will be given.
  Interventions: Biological: Hualan Biology ACYW135 meningococcal polysaccharide vaccine
- age of 2-6 years old,experimental (Experimental): 0.5 ml of Tiantan Biology ACYW135 meningococcal polysaccharide vaccine will be given.
  Interventions: Biological: Tiantan Biology ACYW135 meningococcal polysaccharide vaccine
- age of 2-6 years old,control (Active Comparator): 0.5 ml of Hualan Biology ACYW135 meningococcal polysaccharide vaccine will be given.
  Interventions: Biological: Hualan Biology ACYW135 meningococcal polysaccharide vaccine

INTERVENTIONS:
Biological: Tiantan Biology ACYW135 meningococcal polysaccharide vaccine — Tiantan Biology ACYW135 meningococcal polysaccharide vaccine, intramuscular injection, 0.5 ml
  Arms: age of 18-50 years old, experimental; age of 2-6 years old,experimental; age of 7-17 years old,experimental
Biological: Hualan Biology ACYW135 meningococcal polysaccharide vaccine — Hualan Biology ACYW135 meningococcal polysaccharide vaccine, intramuscular injection, 0.5 ml
  Arms: age of 18-50 years old, control; age of 2-6 years old,control; age of 7-17 years old, control

SUMMARY:
This study evaluates the safety and immunogenicity of the ACYW135 Meningococcal Polysaccharide Vaccine in population aged 2-50 years old. Subjects will be divided into 3 group according to their age, receiving the test vaccine and the control vaccine at the proportion of 1:1 randomly. Each age group has 400 subjects, 1200 in total.

ELIGIBILITY:
Inclusion Criteria:

* With the subject (or his guardian's) informed consent and signed the informed consent;
* The history, physical examination and clinical judgement were determined to be healthy and in accordance with the vaccination age of the product;
* The Subject or his guardian could comply with the clinical study protocol;
* Have not been inoculated with Meningococcal vaccine in the past six months and A + C meningococcal polysaccharide vaccine in the past two years;
* Have not been inoculated with other preventive biological products;
* Axillary temperature≤37.0 ℃.

Exclusion Criteria:

* Children with the history of Neisseria meningitis;
* Had allergies or serious adverse reactions of previous vaccination, such as allergies, urticaria, dyspnea, edema, abdominal pain, etc;
* Had immune inhibitor therapy and cytotoxic therapy, inhaled corticosteroids in the past 6 months (not including allergic rhinitis corticosteroid aerosol therapy, patients with acute non concurrent dermatitis surface corticosteroid therapy);
* Have been accepted blood products in the past 3 months;
* Have been inoculated with other research drugs or vaccines in the past month;
* Have been inoculated with attenuated live vaccine in the past 14 days;
* Have been inoculated with subunit or inactivated vaccine in the past 7 days;
* Had any acute illness, the need for systemic application of antibiotics or antiviral treatment in the past 7 days;
* Had fever in the past 3 days (axillary temperature≥38.0℃) ;
* Have been diagnosed with abnormal coagulation function (such as the lack of coagulation factors, coagulation disorders and abnormal blood platelet), obvious bruises or coagulation disorders by physician diagnosis;
* Had the history of thyroid resection or the need for treatment of thyroid diseases in the past 12 months;
* Asplenia, functional asplenia and asplenia or splenectomy of any situation;
* Had epilepsy, convulsions, encephalopathy, mental illness or family history;
* Suffering from serious chronic diseases (such as Down's syndrome, diabetes, sickle cell anemia, neurological disorders or Guillain-Barre syndrome);
* Suffering from known or suspected concurrent diseases including: respiratory diseases, acute or chronic infection of the activities, children's mother or the subject had HIV infection, cardiovascular disease, high blood pressure, during cancer treatment period, skin diseases;
* The female during her pregnant and lactation period or who plan to become pregnant during the trial.
* The subject of any other factors that are not suitable to participate in clinical trials according to the researcher's judgment.

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1200 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate serum antibody titers of quadrivalent influenza Vaccine in healthy people. | 28 days
  The serum antibody titers will be evaluated at 28 days after vaccination.
Evaluate the Rate of Adverse reactions of quadrivalent influenza Vaccine in healthy people. | 28 days
  Adverse reactions associated with vaccine will be observed in subjects after vaccination. Solicited local adverse events include Pain, Redness, Swelling, Induration, Rash, Pruritus at injection site. solicited general adverse events include Fever, Nausea, Vomiting, Diarrhea, Decreased appetite, Be agitated (irritability, abnormal crying), fatigue, allergy.